CLINICAL TRIAL: NCT01267136
Title: A Comparison of Postoperative Tramadol Versus Acetaminophen With Codeine in Children Undergoing Tonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1010-086
Record Dates: First submitted 2010-12-23; First posted 2010-12-28 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Tonsillitis; Pain
Keywords: Tonsillectomy; Pain; Pediatric; Opioids; Tramadol; Codeine
MeSH Terms: conditions — Tonsillitis; Pain | interventions — Codeine; Acetaminophen; Economics; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capital® with Codeine Suspension (Experimental)
  Interventions: Drug: Codeine with acetaminophen
- Tramadol suspension (Active Comparator)
  Interventions: Drug: Tramadol suspension

INTERVENTIONS:
Drug: Codeine with acetaminophen — Liquid codeine/acetaminophen (Capital® 5mL= 120mg acetaminophen/12 mg codeine) 0.72 mg/kg [=0.3 mL/kg] (max. 36 mg) PO Q6h, plus 0.72 mg/kg (max. 36 mg) PO Q3h pro re nata (PRN) (max. of 3 PRN doses/day)
  Other Names: Capital® with Codeine Suspension; Acetaminophen and Codeine phosphate suspension
  Arms: Capital® with Codeine Suspension
Drug: Tramadol suspension — Liquid tramadol 1.05 mg/kg [=0.3 mL/kg] (max. 52.5 mg) PO Q6h, plus 1.05 mg/kg (max. 52.5 mg) PO Q3h PRN (max. of 3 PRN doses/day).
  Other Names: tramadol hydrochloride; Ultram
  Arms: Tramadol suspension

SUMMARY:
Tonsillectomy is the most common pediatric surgical procedure performed in the US. The postoperative period can be particularly painful. Codeine (usually in mixed formulation with acetaminophen) is the most commonly prescribed opioid in the US. However, evolving data questions its ability to provide optimal pain relief, while avoiding side effects, especially in the postoperative setting. Tramadol may be a better option for children in the postoperative setting due to its well-documented analgesic properties, low potential for side effects, and excellent safety profile. Seventy-two children scheduled to undergo tonsillectomy (with or without adenoidectomy) at Children's will be invited to participate in a randomized, prospective, double-blinded study to evaluate the efficacy and side effects of codeine with acetaminophen versus tramadol. Using a 10-day take-home diary, caregivers will be asked to record daily information about their child's postoperative pain and other core outcomes and domains as recommended in the recent consensus statement put forth by the Pediatric Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) (McGrath et al., 2008). This study will offer new information regarding the efficacy and side effects associated with tramadol as compared with codeine/acetaminophen (the current practice standard) in a pediatric population.

Hypotheses

H1: Children who receive scheduled tramadol following tonsillectomy will report better pain control than children who receive scheduled codeine/acetaminophen.

H2: Children who receive scheduled tramadol following tonsillectomy will report fewer side effects than children who receive scheduled codeine/acetaminophen.

ELIGIBILITY:
Inclusion Criteria:

* Child must be scheduled to undergo tonsillectomy (with or without adenoidectomy).
* Child must be between the ages of 4 and 15 at the time of enrollment.
* Child and caregiver must be English-speaking.
* The same caregiver (e.g., mother) must agree to complete all study assessments with child to ensure consistency.

Exclusion Criteria:

* Child cannot self-assess pain due to conditions such as developmental delays, chromosomal abnormalities, and other syndromes.
* Child had significant adverse effects to codeine, tramadol, or acetaminophen in the past.
* Child has a known underlying seizure disorder (not febrile seizure).
* Child has known underlying renal or liver dysfunction (with creatinine, aspartate aminotransferase [AST]/amino alanine transferase [ALT], above normal value for age, respectively).
* Child or caregiver is not English-speaking.
* The same caregiver (e.g., mother) is unable to complete all follow-up assessments.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Friedrichsdorf, M.D., Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Atef A, Fawaz AA. Peritonsillar infiltration with tramadol improves pediatric tonsillectomy pain. Eur Arch Otorhinolaryngol. 2008 May;265(5):571-4. doi: 10.1007/s00405-007-0479-6. Epub 2007 Oct 17. PMID 17940786
- [Background] Bamigbade TA, Langford RM. Tramadol hydrochloride: an overview of current use. Hosp Med. 1998 May;59(5):373-6. PMID 9722388
- [Background] Chambers CT, Finley AG, McGrath PJ, Walsh TM. The parents' postoperative pain measure: replication and extension to 2-6-year-old children. Pain. 2003 Oct;105(3):437-443. doi: 10.1016/S0304-3959(03)00256-2. PMID 14527704
- [Background] Chambers CT, Reid GJ, McGrath PJ, Finley GA. Development and preliminary validation of a postoperative pain measure for parents. Pain. 1996 Dec;68(2-3):307-13. doi: 10.1016/s0304-3959(96)03209-5. PMID 9121819
- [Background] Chu YC, Lin SM, Hsieh YC, Chan KH, Tsou MY. Intraoperative administration of tramadol for postoperative nurse-controlled analgesia resulted in earlier awakening and less sedation than morphine in children after cardiac surgery. Anesth Analg. 2006 Jun;102(6):1668-73. doi: 10.1213/01.ANE.0000219587.02263.A0. PMID 16717306
- [Background] Ciszkowski C, Madadi P, Phillips MS, Lauwers AE, Koren G. Codeine, ultrarapid-metabolism genotype, and postoperative death. N Engl J Med. 2009 Aug 20;361(8):827-8. doi: 10.1056/NEJMc0904266. No abstract available. PMID 19692698
- [Background] Clark E, Plint AC, Correll R, Gaboury I, Passi B. A randomized, controlled trial of acetaminophen, ibuprofen, and codeine for acute pain relief in children with musculoskeletal trauma. Pediatrics. 2007 Mar;119(3):460-7. doi: 10.1542/peds.2006-1347. PMID 17332198
- [Background] Desmeules JA. The tramadol option. Eur J Pain. 2000;4 Suppl A:15-21. PMID 11310478
- [Background] Dorn MT FN, Quinn FB. Tonsillitis, Tonsillectomy, and Adenoidectomy. Grand Rounds, UTMB - Department of Otolaryngology. December 1999.
- [Background] Drake A CM. Tonsillectomy. EMedicine2003. Available at: http://www.emedicine.com/ent/topic315.htm.
- [Background] Drendel AL, Gorelick MH, Weisman SJ, Lyon R, Brousseau DC, Kim MK. A randomized clinical trial of ibuprofen versus acetaminophen with codeine for acute pediatric arm fracture pain. Ann Emerg Med. 2009 Oct;54(4):553-60. doi: 10.1016/j.annemergmed.2009.06.005. Epub 2009 Aug 19. PMID 19692147
- [Background] Engelhardt T, Steel E, Johnston G, Veitch DY. Tramadol for pain relief in children undergoing tonsillectomy: a comparison with morphine. Paediatr Anaesth. 2003 Mar;13(3):249-52. doi: 10.1046/j.1460-9592.2003.00983.x. PMID 12641688
- [Background] Finkel JC, Rose JB, Schmitz ML, Birmingham PK, Ulma GA, Gunter JB, Cnaan A, Cote CJ, Medve RA, Schreiner MS. An evaluation of the efficacy and tolerability of oral tramadol hydrochloride tablets for the treatment of postsurgical pain in children. Anesth Analg. 2002 Jun;94(6):1469-73, table of contents. doi: 10.1097/00000539-200206000-00017. PMID 12032009
- [Background] Fortier MM, J; Martin, S; Kain, Z. Children's pain at home following ambulatory surgery. J Pain2009;10(4 (Suppl1)):106.
- [Background] Hain RD, Miser A, Devins M, Wallace WH. Strong opioids in pediatric palliative medicine. Paediatr Drugs. 2005;7(1):1-9. doi: 10.2165/00148581-200507010-00001. PMID 15777107
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Hullett BJ, Chambers NA, Pascoe EM, Johnson C. Tramadol vs morphine during adenotonsillectomy for obstructive sleep apnea in children. Paediatr Anaesth. 2006 Jun;16(6):648-53. doi: 10.1111/j.1460-9592.2005.01827.x. PMID 16719881
- [Background] Marquardt KA, Alsop JA, Albertson TE. Tramadol exposures reported to statewide poison control system. Ann Pharmacother. 2005 Jun;39(6):1039-44. doi: 10.1345/aph.1E577. Epub 2005 May 3. PMID 15870139
- [Background] McGrath PA, Seifert CE, Speechley KN, Booth JC, Stitt L, Gibson MC. A new analogue scale for assessing children's pain: an initial validation study. Pain. 1996 Mar;64(3):435-443. doi: 10.1016/0304-3959(95)00171-9. PMID 8783307
- [Background] McGrath PJ, Walco GA, Turk DC, Dworkin RH, Brown MT, Davidson K, Eccleston C, Finley GA, Goldschneider K, Haverkos L, Hertz SH, Ljungman G, Palermo T, Rappaport BA, Rhodes T, Schechter N, Scott J, Sethna N, Svensson OK, Stinson J, von Baeyer CL, Walker L, Weisman S, White RE, Zajicek A, Zeltzer L; PedIMMPACT. Core outcome domains and measures for pediatric acute and chronic/recurrent pain clinical trials: PedIMMPACT recommendations. J Pain. 2008 Sep;9(9):771-83. doi: 10.1016/j.jpain.2008.04.007. Epub 2008 Jun 17. PMID 18562251
- [Background] McLellan RA, Oscarson M, Seidegard J, Evans DA, Ingelman-Sundberg M. Frequent occurrence of CYP2D6 gene duplication in Saudi Arabians. Pharmacogenetics. 1997 Jun;7(3):187-91. doi: 10.1097/00008571-199706000-00003. PMID 9241658
- [Background] Moir MS, Bair E, Shinnick P, Messner A. Acetaminophen versus acetaminophen with codeine after pediatric tonsillectomy. Laryngoscope. 2000 Nov;110(11):1824-7. doi: 10.1097/00005537-200011000-00011. PMID 11081593
- [Background] Moore A, Collins S, Carroll D, McQuay H. Paracetamol with and without codeine in acute pain: a quantitative systematic review. Pain. 1997 Apr;70(2-3):193-201. doi: 10.1016/s0304-3959(96)03319-2. PMID 9150293
- [Background] Moore AR, McQuay JH. Single-patient data meta-analysis of 3453 postoperative patients: oral tramadol versus placebo, codeine and combination analgesics. Pain. 1997 Feb;69(3):287-294. doi: 10.1016/S0304-3959(96)03291-5. PMID 9085303
- [Background] Nunez DA, Provan J, Crawford M. Postoperative tonsillectomy pain in pediatric patients: electrocautery (hot) vs cold dissection and snare tonsillectomy--a randomized trial. Arch Otolaryngol Head Neck Surg. 2000 Jul;126(7):837-41. doi: 10.1001/archotol.126.7.837. PMID 10888995
- [Background] Oxford Pain Site. Available at: http://www.medicine.oc.ac.uk/bandolier/booth/painpag/acute.html
- [Background] Pendeville PE, Von Montigny S, Dort JP, Veyckemans F. Double-blind randomized study of tramadol vs. paracetamol in analgesia after day-case tonsillectomy in children. Eur J Anaesthesiol. 2000 Sep;17(9):576-82. doi: 10.1046/j.1365-2346.2000.00729.x. PMID 11029125
- [Background] Rose JB, Finkel JC, Arquedas-Mohs A, Himelstein BP, Schreiner M, Medve RA. Oral tramadol for the treatment of pain of 7-30 days' duration in children. Anesth Analg. 2003 Jan;96(1):78-81, table of contents. doi: 10.1097/00000539-200301000-00016. PMID 12505927
- [Background] Sidman JD, Lander TA, Finkelstein M. Platelet-rich plasma for pediatric tonsillectomy patients. Laryngoscope. 2008 Oct;118(10):1765-7. doi: 10.1097/MLG.0b013e31817f18e7. PMID 18622315
- [Background] Sutters KA, Miaskowski C, Holdridge-Zeuner D, Waite S, Paul SM, Savedra MC, Lanier B. Time-contingent dosing of an opioid analgesic after tonsillectomy does not increase moderate-to-severe side effects in children. Pain Manag Nurs. 2005 Jun;6(2):49-57. doi: 10.1016/j.pmn.2005.01.001. PMID 15970918
- [Background] von Baeyer CL, Spagrud LJ, McCormick JC, Choo E, Neville K, Connelly MA. Three new datasets supporting use of the Numerical Rating Scale (NRS-11) for children's self-reports of pain intensity. Pain. 2009 Jun;143(3):223-227. doi: 10.1016/j.pain.2009.03.002. Epub 2009 Apr 8. PMID 19359097
- [Background] Williams DG, Patel A, Howard RF. Pharmacogenetics of codeine metabolism in an urban population of children and its implications for analgesic reliability. Br J Anaesth. 2002 Dec;89(6):839-45. doi: 10.1093/bja/aef284. PMID 12453926

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was introduced to 137 potential subjects during or following an outpatient office evaluation with an ear/nose/throat (ENT) surgeon between February 2011 and May 2012.
Pre-assignment Details: The study was introduced to 137 potential subjects, and 84 children were enrolled in the study and assigned to one of the two study arms.
Groups:
- Capital® With Codeine Suspension: Codeine with acetaminophen : Liquid codeine/acetaminophen (Capital® 5mL= 120mg acetaminophen/12 mg codeine) 0.72 mg/kg [=0.3 mL/kg] (max. 36 mg) PO Q6h, plus 0.72 mg/kg (max. 36 mg) PO Q3h pro re nata (PRN) (max. of 3 PRN doses/day)
- Tramadol Suspension: Tramadol suspension : Liquid tramadol 1.05 mg/kg [=0.3 mL/kg] (max. 52.5 mg) PO Q6h, plus 1.05 mg/kg (max. 52.5 mg) PO Q3h pro re nata (PRN) (max. of 3 PRN doses/day).
Period: Overall Study
Arm/Group | Capital® With Codeine Suspension | Tramadol Suspension
Started | 42 | 42
Completed | 38 | 36
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Capital® With Codeine Suspension: Codeine with acetaminophen : Liquid codeine/acetaminophen (Capital® 5mL= 120mg acetaminophen/12 mg codeine) 0.72 mg/kg [=0.3 mL/kg] (max. 36 mg) PO Q6h, plus 0.72 mg/kg (max. 36 mg) PO Q3h PRN (max. of 3 PRN doses/day)
- Tramadol Suspension: Tramadol suspension : Liquid tramadol 1.05 mg/kg [=0.3 mL/kg] (max. 52.5 mg) PO Q6h, plus 1.05 mg/kg (max. 52.5 mg) PO Q3h PRN (max. of 3 PRN doses/day).
- Total: Total of all reporting groups
Arm/Group | Capital® With Codeine Suspension | Tramadol Suspension | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 42 | 84
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.4 (2.3) | 6.6 (2.3) | 6.5 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 16 | 17 | 33
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Two Different Liquid Pain Medications: Tramadol vs. Codeine/Acetaminophen During the Post-tonsillectomy Recovery Period.
Description: Average number of post-operative days with pain score >4/10. Pain score assessments were administered once daily by parents using either the Numeric Rating Scale (NRS-11) (with anchors 0=no pain and 10=highest pain imaginable) for children ages 8-15 (von Baeyer et al., 2009) or the Faces Pain Scale-Revised (FPS-R) (with anchors 0=no pain and 10=highest pain imaginable) for children ages 4-10 (Hicks et al., 2001).
Time Frame: Efficacy was assessed daily during the 10-day postoperative recovery period.
Measure: Median (Full Range); unit: days
Arm/Group | Capital® With Codeine Suspension | Tramadol Suspension
Number analyzed (Participants) | 38 | 36
days | 1.5 [0 to 9] | 1 [0 to 9]

2. Secondary Outcome: Number of Participants Reporting Side Effects During the Post-tonsillectomy Recovery Period.
Description: Parent-reported side effects entered in 10-day diary.
Time Frame: Side effects will be observed and recorded daily by caregivers for a total of 10 days in the take-home diary.
Measure: Number; unit: participants
Groups:
- Capital® With Codeine Suspension: Codeine with acetaminophen: Liquid codeine/acetaminophen (Capital® 5mL= 120mg acetaminophen/12 mg codeine) 0.72 mg/kg [=0.3 mL/kg] (max. 36 mg) PO Q6h, plus 0.72 mg/kg (max. 36 mg) PO Q3h PRN (max. of 3 PRN doses/day)
Arm/Group | Capital® With Codeine Suspension | Tramadol Suspension
Number analyzed (Participants) | 38 | 36
participants
  Nausea | 20 | 20
  Vomiting | 21 | 18
  Fever | 11 | 10
  Itching | 5 | 12
  Rash | 1 | 1
  Sweating | 9 | 7
  Dizziness | 15 | 17
  Headache | 12 | 17
  Constipation | 21 | 21
  Oversedation | 14 | 8
  Tonsil bleed | 3 | 0

ADVERSE EVENTS:
Arm/Group | Capital® With Codeine Suspension | Tramadol Suspension
Serious Adverse Events (participants affected / at risk) | 1/42 | 1/42
Other Adverse Events (participants affected / at risk) | 33/38 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capital® With Codeine Suspension (N=42) | Tramadol Suspension (N=42)
Tonsil bleed requiring hospitalization (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Patient had hypoplastic left heart syndrome and was pacemaker-dependent. This child experienced a life-threatening tonsil hemorrhage one week after surgery, requiring resuscitation and hospitalization, and discontinuation of the study medication.
Throat pain requiring hospitalization (General disorders) | 0 (0) | 1 (1) — Patient was hospitalized for difficulty with oral intake, dehydration, and throat pain. This patient was rehydrated and switched to acetaminophen and hydrocodone (Lortab) for pain management following discharge.
Dehydration (General disorders) | 0 (0) | 1 (1) — Patient was hospitalized for difficulty with oral intake, dehydration, and throat pain. This patients was rehydrated and switched to acetaminophen and hydrocodone (Lortab) for pain management following discharge.
Difficulty with oral intake (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient was hospitalized for difficulty with oral intake, dehydration, and throat pain. This patients was rehydrated and switched to acetaminophen and hydrocodone (Lortab) for pain management following discharge.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capital® With Codeine Suspension (N=38) | Tramadol Suspension (N=36)
Nausea (Nervous system disorders) | 20 | 20
Vomiting (Gastrointestinal disorders) | 21 | 18
Fever (Infections and infestations) | 11 | 10
Itching (Skin and subcutaneous tissue disorders) | 5 | 12
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Sweating (General disorders) | 9 | 7
Dizziness (Nervous system disorders) | 15 | 17
Headache (Nervous system disorders) | 12 | 17
Constipation (Gastrointestinal disorders) | 21 | 21
Oversedation (General disorders) | 14 | 8
Tonsil bleed (Blood and lymphatic system disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
There was insufficient power to detect differences in safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No